CLINICAL TRIAL: NCT00587769
Title: Combination Pharmacotherapy With Chantix & Bupropion for Smoking Cessation (ChanBan)
Brief Title: Chantix & Bupropion for Smoking Cessation
Acronym: ChanBan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jon Ebbert, Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-003998
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Smoking; Tobacco Use Disorder
Keywords: Smoking; Smoking cessation; Bupropion; Varenicline; Tobacco use disorder
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion SR & Varenicline (Experimental): All 38 smokers will receive open-label bupropion SR and varenicline. Bupropion SR is an oral medication with recommended dosing of 150 mg by mouth once day for 3 days then 150 mg by mouth twice per day. Varenicline is an oral medication with recommended dosing of 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4 to 7, and then to the maintenance dose of 1 mg twice daily for the 12 weeks of treatment. Subjects will quit on Day #8 after starting both medications.
  Interventions: Drug: Bupropion SR & Varenicline

INTERVENTIONS:
Drug: Bupropion SR & Varenicline — Bupropion SR 150 mg by mouth once day for 3 days then 150 mg by mouth twice per day.
  Varenicline 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4 to 7, and then to the maintenance dose of 1 mg twice daily for the 12 weeks of treatment.

SUMMARY:
The overarching goal of this line of research is to increase smoking abstinence rates using a combination of existing pharmacotherapies. The aim of the current study is to assess the safety and compliance as well as obtain preliminary estimates of efficacy and effect on craving and nicotine withdrawal of combination therapy with bupropion SR and varenicline. We will compare the efficacy estimates in this study with historical smoking abstinence rates with varenicline. To accomplish our aims, we will enroll 38 cigarette smokers in an open-label, phase II clinical trial.

DETAILED DESCRIPTION:
Subjects will be eligible to participate if they: 1) are at least 18 years of age; 2) have smoked 10 or more cigarettes per day for at least 6 months; and 3) are motivated to stop smoking.

Subjects will be excluded if they have: 1) an unstable medical condition; 2) unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months or an untreated cardiac dysrhythmia; 3) personal history of seizures; 4) closed head trauma with any loss of consciousness or amnesia in the last 5 years; 5) ever history of closed head trauma with > 30 minutes of loss of consciousness or amnesia or resulting in skull fracture or subdural hematoma/brain contusion; 6) a history or psychosis, bipolar disorder, bulimia or anorexia nervosa); 7) have current depression as assessed by Center for Epidemiologic Studies Depression (CES-D); 8) have active substance abuse other than nicotine; 9) have used an investigational drug within the last 30 days; 10) are currently using a behavioral or pharmacologic tobacco treatment and unwilling or unable to discontinue use; 11) use of bupropion or varenicline in the previous 3 months; 12) current (past 14 days) use of antipsychotic or antidepressant; 13) an allergy to bupropion or varenicline; 14) untreated hypertension or baseline systolic blood pressure > 180 or diastolic > 100; 15) have another member of their household already participating in this study.

The primary aims and hypotheses of this study are:

1. To obtain preliminary evidence of efficacy of 12 weeks of combination therapy with bupropion SR and varenicline for increasing the point prevalence smoking abstinence rates at 12 weeks among cigarette smokers.

   Hypothesis: The combination of bupropion SR plus varenicline for 12 weeks will increase the point prevalence smoking abstinence rates at 12 weeks among cigarettes smokers.
2. To obtain preliminary evidence of efficacy of combination therapy with bupropion SR and varenicline for decreasing craving and nicotine withdrawal symptoms among cigarette smokers trying to achieve smoking abstinence.

Hypothesis: 12 weeks of combination therapy with bupropion SR and varenicline will significantly decrease craving and nicotine withdrawal among cigarette smokers trying to achieve smoking abstinence.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* have smoked 10 or more cigarettes per day for at least 6 months
* are motivated to stop smoking.

Exclusion Criteria:

* an unstable medical condition
* unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months or an untreated cardiac dysrhythmia
* personal history of seizures
* closed head trauma with any loss of consciousness or amnesia in the last 5 years
* ever history of closed head trauma with > 30 minutes of loss of consciousness or amnesia or resulting in skull fracture or subdural hematoma/brain contusion
* a history or psychosis, bipolar disorder, bulimia or anorexia nervosa)
* have current depression as assessed by Center for Epidemiologic Studies Depression (CES-D)
* have active substance abuse other than nicotine
* have used an investigational drug within the last 30 days
* are currently using a behavioral or pharmacologic tobacco treatment and unwilling or unable to discontinue use
* use of bupropion or varenicline in the previous 3 months
* current (past 14 days) use of antipsychotic or antidepressant
* an allergy to bupropion or varenicline
* untreated hypertension or baseline systolic blood pressure > 180 or diastolic > 100
* have another member of their household already participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O Ebbert, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Nicotine Research Program — http://ndc.mayo.edu/mayo/research/nicotine_research_center/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient's were recruited between 10 September, 2007 and 25 October, 2007 in the community surrounding the Mayo Clinic in Rochester Minnesota.
Pre-assignment Details: Patients were excluded for not meeting entry criteria
Groups:
- Medication Arm: Varenicline 1.0 mg po bid plus bupropion 150 mg po bid
Period: Overall Study
Arm/Group | Medication Arm
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medication Arm
Number analyzed (Participants) | 38
Age Continuous [Median (Standard Deviation); unit: years] | 49.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 19.9 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Smoking Abstinence at 12 Weeks: the Number of Patients Who Refrained From Smoking at 12 Weeks
Description: Smoking abstinence biochemically confirmed with exhaled carbon monoxide concentrations
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Medication Arm
Number analyzed (Participants) | 38
Participants | 27 [54 to 85]

2. Secondary Outcome: Point Prevalence Smoking Abstinence at 6 Months: the Number of Patients Who Refrained From Smoking at 6 Months
Description: Smoking abstinence biochemically confirmed with exhaled carbon monoxide concentrations
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Medication Arm
Number analyzed (Participants) | 38
Participants | 22

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Medication Arm
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 25/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Arm (N=38)
Sleep disturbance (Nervous system disorders) | 10 (10)
Nausea (Nervous system disorders) | 9 (9)
Insomnia (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5)
Vivid dreams (Nervous system disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Dry mouth (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No